CLINICAL TRIAL: NCT00636311
Title: IGEV +/- Bortezomib (Velcade) as Induction Before High Dose Consolidation in Relapsed/Refractory Hodgkin's Lymphoma After First Line Treatment: a Randomized Phase II Trial. On Behalf of Intergruppo Italiano Linfomi
Brief Title: A Phase II Study of IGEV +/- Bortezomib Before Hign Dose Consolidation in Relapsed/Refractory Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Armando Santoro, MD, Istituto Clinico Humanitas
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ONC-2006-005; EUDRACT 2007-004883-29
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2010-09-02 (Estimated); Status verified 2010-09

CONDITIONS: Hodgkin Disease
Keywords: Hodgkin disease; Salvage therapy; Bortezomib; Transplantation
MeSH Terms: conditions — Hodgkin Disease | interventions — Ifosfamide; Gemcitabine; Vinorelbine; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): IGEV regimen (Ifosfamide, Gemcitabine, Vinorelbine)
  Interventions: Drug: Ifosfamide, Gemcitabine, Vinorelbine
- 2 (Experimental): B-IGEV (Bortezomib + IGEV)
  Interventions: Drug: Bortezomib + IGEV

INTERVENTIONS:
Drug: Ifosfamide, Gemcitabine, Vinorelbine — Ifosfamide 2000 mg/sqm, day 1-4 (plus MESNA); Gemcitabine 800 mg/sqm, day 1 and 4; Vinorelbine 20 mg/sqm, day 1; Prednisone 100 mg, day 1-4; G-CSF 1 vial sc, day 7-12 of each 21-day course.
  Arms: 1
Drug: Bortezomib + IGEV — Bortezomib 1,3 mg/sqm, day 1, 4, 8; Ifosfamide 2000 mg/sqm, day 1-4 (plus MESNA); Gemcitabine 800 mg/sqm, day 1 and 4; Vinorelbine 20 mg/sqm, day 1; Prednisone 100 mg, day 1-4; G-CSF 1 vial sc, day 7-12 of each 21-day course.
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate if the addition of Bortezomib (Velcade) to IGEV combination (Ifosfamide, Gemcitabine and Vinorelbine) in patients with relapsed/refractory Hodgkin's lymphoma increases the rate of complete remission (PET negativity) at transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Hodgkin's lymphoma failing or relapsing after first-line chemotherapy (MOPP/AVBD , MOPP/EBV/CAD and analogs are considered one line)
* Age >18 and <65 years
* Signed informed consent
* If female, patient is either postmenopausal or surgically sterilized or willing to use an acceptable method of birth control
* If male, patient agrees to use an acceptable barrier method for contraception
* ECOG performance status <2
* Platelet count >100.000/mmc
* Hemoglobin >7.5 g/dL
* Absolute neutrophil count (ANC) >1.500/mmc
* Serum calcium <3.5 mmol/L (<14 mg/dL)
* AST/ALT: <2.5 x the ULN
* Total bilirubin: <1.5 x the ULN

Exclusion Criteria:

* Previous treatment with velcade
* Nitrosoureas within 6 weeks or any other chemotherapy within 3 weeks before enrollment
* Immunotherapy or antibody therapy within 4 weeks before enrollment
* Experimental drug or medical device within 4 weeks before start of treatment
* Major surgery within 4 weeks before enrollment
* History of allergic reaction attributable to compounds containing boron or mannitol or any of the drugs in the IGEV regimen
* Peripheral neuropathy of NCI CTCAE Grade 2 or higher
* Myocardial infarction within 6 months of enrollment or NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* History of clinically relevant liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, rheumatologic, hematologic, psychiatric, or metabolic disturbances including diabetes mellitus
* Need for therapy with concomitant CYP 3A4 inhibitors or inducers
* HIV-positive, if known
* Hepatitis B surface antigen-positive or active hepatitis C infection, if known
* Active systemic infection requiring treatment
* If female, pregnancy or breast-feeding.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-02; Primary Completion 2008-04 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
PET negativity rate obtained with IGEV or B-IGEV will be compared | PET negativity after 4 courses of induction (IGEV or B-IGEV)

CONTACTS AND LOCATIONS:
Overall Officials: Armando Santoro, MD, Principal Investigator — Istituto Clinico Humanitas
Locations (1):
- Istituto Clinico Humanitas, Rozzano, Milan, Italy

REFERENCES:
- [Background] Santoro A, Magagnoli M, Spina M, Pinotti G, Siracusano L, Michieli M, Nozza A, Sarina B, Morenghi E, Castagna L, Tirelli U, Balzarotti M. Ifosfamide, gemcitabine, and vinorelbine: a new induction regimen for refractory and relapsed Hodgkin's lymphoma. Haematologica. 2007 Jan;92(1):35-41. doi: 10.3324/haematol.10661. PMID 17229633